CLINICAL TRIAL: NCT06659445
Title: A Phase 2 Multicenter, Randomized, Double-masked, Sham-controlled, Reference-arm Study to Evaluate Efficacy and Safety of ONL1204 in Patients With Geographic Atrophy (GA) Associated With Age-related Macular Degeneration (AMD)
Brief Title: Study to Evaluate Efficacy and Safety of ONL1204 in Patients With GA Associated With AMD
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: ONL Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ONL1204-GA-002
Record Dates: First submitted 2024-10-23; First posted 2024-10-26 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Geographic Atrophy (GA); Age - Related Macular Degeneration (AMD)
Keywords: Phase 2; ONL1204; Geographic Atrophy (GA); Age-related Macular Degeneration (AMD)
MeSH Terms: conditions — Geographic Atrophy; Macular Degeneration | interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- ONL1204 Opthalmic solution (1 of 6 Treatment Groups) administered by intravitreal injection (Active Comparator): ONL1204 100 µg administered by intravitreal (IVT) injection every 12 weeks
  Interventions: Drug: ONL1204 Opthalmic solution
- ONL1204 Opthalmic solution (2 of 6 Treatment Groups) administered by intravitreal injection (Active Comparator): ONL1204 200 µg administered by intravitreal (IVT) injection every 12 weeks
  Interventions: Drug: ONL1204 Opthalmic solution
- ONL1204 Opthalmic solution (3 of 6 Treatment Groups) administered by intravitreal injection (Experimental): ONL1204 200 µg administered by intravitreal (IVT) injection every 24 weeks
  Interventions: Drug: ONL1204 Opthalmic solution
- Sham Comparator (4 of 6 Treatment Groups) (Sham Comparator): Sham injection every 12 weeks
  Interventions: Other: Sham
- Sham Comparator (5 of 6 Treatment Groups) (Sham Comparator): Sham injection every 24 weeks
  Interventions: Other: Sham
- Avacincaptad pegol intravitreal solution (6 of 6 Treatment Groups - US ONLY) (Active Comparator): Avacincaptad pegol administered by intravitreal (IVT) injection - (2 mg (0.1 mL of 20 mg/mL solution) once monthly
  Interventions: Drug: Avacincaptad Pegol intravitreal solution

INTERVENTIONS:
Drug: ONL1204 Opthalmic solution — Liquid formulation ONL1204 Ophthalmic Solution administered by intravitreal (IVT) injection
  Arms: ONL1204 Opthalmic solution (1 of 6 Treatment Groups) administered by intravitreal injection; ONL1204 Opthalmic solution (2 of 6 Treatment Groups) administered by intravitreal injection; ONL1204 Opthalmic solution (3 of 6 Treatment Groups) administered by intravitreal injection
Drug: Avacincaptad Pegol intravitreal solution — Liquid formulation Avacincaptad Pegol administered by intravitreal (IVT) injection
  Arms: Avacincaptad pegol intravitreal solution (6 of 6 Treatment Groups - US ONLY)
Other: Sham — Sham injection
  Arms: Sham Comparator (4 of 6 Treatment Groups); Sham Comparator (5 of 6 Treatment Groups)

SUMMARY:
The purpose of this study is to collect efficacy and safety information of intravitreal injection for 3 experimental arms, including 2 dose levels of ONL1204 and 2 treatment frequencies in patients with GA associated with AMD.

GA associated with AMD is one of the world's leading causes of visual disability and legal blindness globally. Associated with aging, cigarette smoking, obesity, diets low in certain nutrients, a lifestyle related to cardiac risk, and a growing list of genetic factors, AMD is becoming an increasingly prevalent public health concern, especially as the global population ages. ONL1204 is a first-in-class inhibitor of fragment apoptosis stimulator receptor-mediated cell death that has demonstrated protection of multiple retinal cell types in numerous preclinical models of retinal disease, including models of dry AMD.

ELIGIBILITY:
Inclusion Criteria:

1. 55 years of age or older at Screening.
2. Able and willing to give informed consent and attend study visits.
3. Women or intersex individuals must be willing to use 2 forms of effective contraception during the study and for at least 90 days following the last dose of study drug, be postmenopausal for at least 12 months prior to study entry, or surgically sterile. If of childbearing potential, a negative urine pregnancy test is required at Screening and prior to the administration of study drug at each visit.
4. Men or intersex individuals with partners of childbearing potential must be willing to use permissible methods of contraception and refrain from sperm donation during the study and for at least 90 days following the last dose of study drug.
5. If currently using Age-related Eye Disease Study 2 (AREDS, AREDS2, or similar nutraceutical therapy at Screening, patient must be willing to continue use for the duration of the study. If not currently using AREDS2 or similar, patient must be willing to continue not to use therapy for the duration of the study. Patient must agree to choose either approach.

   Study Eye Inclusion Criteria:
6. BCVA of 24 letters or more using ETDRS charts in the study eye at Screening.
7. Intraocular pressure (IOP) of 22 mmHg or lower in the study eye at Screening.

   The GA lesion must meet all the following criteria:
8. Non-foveal GA associated with AMD without eMNV in the study eye per Investigator's evaluation and as confirmed by the central RC.
9. GA ≥0.85 disc area (DA) (2.125 mm2) and ≤8.05 DA (20.125 mm2) in the study eye as confirmed by the central RC.
10. If GA in the study eye is multifocal, at least 1 focal lesion must be ≥0.425 DA (1.063 mm2) as confirmed by the central RC.
11. Non-foveal GA (GA lesion up to the fovea, but not subfoveal) with the lesion's closest border 1725 microns or less from the foveal center in the study eye, as confirmed by the central RC.
12. The entire GA lesion in the study eye must be completely visualized on the macula-centered FAF image, must be able to be imaged in its entirety, and must not be contiguous with any areas of peripapillary atrophy per the Investigator's evaluation and as confirmed by the central RC.
13. A pattern of hyper-autofluorescence in the junctional zone of GA in the study eye must be present as confirmed by the central RC.

    Fellow Eye Inclusion Criterion:
14. BCVA of 19 letters or more using ETDRS charts in the fellow eye at Screening.

Exclusion Criteria:

1. Current or planned participation in another investigational clinical study or use of any other investigational drugs or devices at least 6 months prior to enrollment or during the study period without prior written Sponsor approval.
2. Previous ophthalmic disease gene therapy or planned participation in any gene therapy clinical study during the study period.
3. Current or planned use of systemic complement inhibitors during the study period.
4. Any ocular or systemic condition that, in the opinion of the Investigator, makes the patient unsuitable for treatment with an investigational drug or that would compromise the safety or efficacy assessments of the study.
5. Treatment with any ocular or systemic medication that is known to be toxic to the lens, retina, or optic nerve (including, but not limited to, aminoglycosides, vancomycin, hydroxychloroquine, interferon, tacrolimus, cisplatin, bis-chloroethyl nitrosourea, carmustine, ethambutol, and tamoxifen) within 90 days prior to Screening or anticipated during the study period.
6. Any previous treatment of pentosan polysulfate (Elmiron®) is exclusionary.
7. Known allergy to fluorescein, povidone iodine, or any ingredients of the study drug or avacincaptad pegol intravitreal solution.
8. Individuals who are currently pregnant, planning to become pregnant, or are nursing at Screening or during the study period.

   Study Eye Exclusion Criteria:
9. Active ocular or periocular infection in the study eye.
10. Any contraindication to an IVT injection in the study eye.
11. Any media opacity in the study eye that limits visual acuity, clinical visualization of the retina, or retinal imaging as determined by the Investigator.
12. Previous IVT pharmaceutical treatment in the study eye with any agent except Food and Drug Administration (FDA)-approved complement inhibitors and treatment with FDA-approved complement inhibitors within 12 weeks prior to Screening.
13. Any history of incisional retinal surgery in the study eye including but not limited to scleral buckle or vitrectomy. (Retinal laser for a tear or hole 3 months or more prior to Screening is not exclusionary).
14. History of incisional glaucoma surgery including trabeculectomy, tube shunt, or minimally invasive glaucoma surgery in the study eye. (Glaucoma laser procedures performed at least 6 months prior to Screening are not exclusionary).
15. Yttrium aluminum garnet capsulotomy in the study eye within 1 month prior to Screening.
16. Cataract surgery in the study eye planned or expected during the study period.
17. Aphakia with absence of the posterior capsule in the study eye. (Pseudophakia with an open posterior capsule is not exclusionary).
18. Any current evidence or history in the study eye of exudative ("wet") AMD, including any RPE rips or evidence of actively leaking neovascularization anywhere in the retina based on the FA or SD-OCT as assessed per the Investigator's evaluation and confirmed by the central RC.
19. Any clinically significant retinal disease other than AMD except benign degenerative conditions (eg, Cobblestone degeneration) in the study eye.
20. Intraocular surgery in the study eye (including lens replacement surgery) within 3 months prior to Screening. See Exclusion Criteria 12 and 13 pertaining to retinal and glaucoma surgery, respectively.
21. Previous therapeutic radiation (including transpupillary thermotherapy, photodynamic therapy, or external-beam) in the region of the study eye.

    Fellow Eye Exclusion Criterion:
22. Planned or expected IVT injection in the fellow eye for treatment of GA with agents other than FDA-approved complement inhibitors (pegcetacoplan or avacincaptad pegol IVT solution [Izervay™]) during the study period.

    Either Eye Exclusion Criteria:
23. Active intraocular inflammation in either eye or a history of uveitis or endophthalmitis in either eye.
24. GA in either eye due to causes other than AMD.
25. Any ophthalmic condition in either eye that is likely to require surgery during the study period.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 324 (Estimated)
Dates: Start 2025-10-28 (Actual); Primary Completion 2028-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Primary Endpoint | From enrollment to the end of treatment at 48 weeks.
  GA lesion area

SECONDARY OUTCOMES:
Secondary Endpoints (Safety) | From enrollment to the end of treatment at 48 weeks.
  Incidence of new active exudative macular neovascularization (eMNV) in the study eye
Secondary Endpoints (Safety) | From enrollment to the end of treatment at 48 weeks.
  Incidence of Early Treatment of Diabetic Retinopathy Study (ETDRS) best corrected visual acuity (BCVA) loss

CONTACTS AND LOCATIONS:
Locations (28):
- United States (27):
  - Associated Retina Consultants, Gilbert, Arizona
  - Associated Retina Consultants, Phoenix, Arizona
  - Doheny Image Reading Center, Pasadena, California
  - Bay Area Retina Associates, Walnut Creek, California
  - Retina Consultants of Southern Colorado, Colorado Springs, Colorado
  - Retina Group of New England, Waterford, Connecticut
  - Florida Retina Institute, Orlando, Florida
  - Retina Associates, Ltd., Elmhurst, Illinois
  - Retina Partners Midwest, P.C., Carmel, Indiana
  - Retina Research Institute at New England Retina Consultants, Springfield, Massachusetts
  - Associated Retinal Consultants, P.C., Royal Oak, Michigan
  - The Retina Institute, St Louis, Missouri
  - Sierra Eye Associates, Reno, Nevada
  - Retina Associates of Western NY, Rochester, New York
  - Long Island Vitreoretinal Consultants, Westbury, New York
  - North Carolina Retina Associates, S.C., Wake Forest, North Carolina
  - Erie Retina Research, LLC (Clinic), Erie, Pennsylvania
  - Charleston Neuroscience Institute, Mt. Pleasant, South Carolina
  - Palmetto Retina Center, West Columbia, South Carolina
  - Retina Consultants of Texas, Beaumont, Texas
  - Retina Consultants of Texas, Bellaire, Texas
  - Retina Consultants of Texas, Katy, Texas
  - Retina Associates of South Texas, PA, San Antonio, Texas
  - Retina Consultants of Texas, San Antonio, Texas
  - Retina Consultants of Texas, The Woodlands, Texas
  - Pacific Northwest Retina, Bellevue, Washington
  - Pacific Northwest Retina, PLLC, Silverdale, Washington
- Clinique d'ophtalmologie des Laurentides, Boisbriand, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes